CLINICAL TRIAL: NCT00674882
Title: Protocol For Collecting Long-Term Follow-Up Data On Recipients of Hematopoietic Stem Cell Transplant
Brief Title: Protocol For Collecting Long-Term Follow-Up Data On Recipients of Bone Marrow and Blood Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BMTFU; NCI-2021-10847 (Registry Identifier: NCI)
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic stem cell transplant; Follow-up studies; Outcomes research; Data collection
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Data Collection
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Data Collection, Outcomes Research, Statistical Data Analysis, Longitudinal Study

SUMMARY:
This protocol allows for ongoing data collection to assess the long-term clinical and psychosocial outcomes of pediatric patients who have received a hematopoietic stem cell transplant at St. Jude Children's Research Hospital.

DETAILED DESCRIPTION:
The purpose of this protocol is to provide ongoing data collection and review of long-term outcome and late effects in a large cohort of St. Jude Children's Research Hospital autologous and allogeneic hematopoietic stem cell recipients. Central coordination of clinical and psychosocial late effects monitoring and reporting can facilitate timely communication about life-threatening or unanticipated clinical outcomes as well as significant psychological, social and behavioral sequelae effects on the recipient and their family members. The resultant data may enable researchers in their development of current clinical and psychosocial studies, as well as monitoring predisposed survivors who may benefit from preventive or corrective interventions. Physicians and researchers may be able to learn how to identify these problems earlier, to take better care of these problems, or to implement preventive measures for future transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* St. Jude patients actively monitored in the BMT-AFU clinic after receiving HSC transplant for a malignant or non-malignant condition.
* St. Jude alumnus who has received a hematopoietic stem cell transplant for a malignant or non-malignant condition and is monitored by the Tumor Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: St. Jude patient at least one year post receipt of an autologous or allogeneic transplant for a malignant or non-malignant condition
Sampling Method: Non-Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
To provide ongoing review of long-term clinical and psychosocial outcomes and late effects of hematopoietic stem cell recipients at St. Jude Children's Research Hospital | Long Term Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols